CLINICAL TRIAL: NCT06133881
Title: A Randomized Comparative Study on the Effect of Using Intrathecal Hyperbaric Prilocaine Plus Fentanyl Compared to Hyperbaric Bupivacaine Plus Fentanyl on the Motor Block in Women Undergoing Caesarean Section Under Spinal Anesthesia
Brief Title: Effect of Prilocaine on Motor Block During Caesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Hassab elnaby, associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MS-268-2023
Record Dates: First submitted 2023-11-02; First posted 2023-11-18 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Spinal for Caesarean Section
Keywords: prilocaine; caesarean section; spinal enesthesia
MeSH Terms: interventions — Prilocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prilocaine (Experimental)
  Interventions: Drug: prilocaine
- bupivacaine (Active Comparator)
  Interventions: Drug: bupivacaine

INTERVENTIONS:
Drug: prilocaine — intrathecal 50 mg (2.5 ml) of prilocaine 2% (Takipril, prilocaine hydrochloride 20 mg/mL, hyperbar, Sintetica) + 25 ug fentanyl (0.5 ml).
  Arms: prilocaine
Drug: bupivacaine — intrathecal 10 mg (2 ml) of bupivacaine 5% (sunnypivacaine hyperbaric bupivacaine 20 mg/4ml + 25 ug fentanyl (0.5 ml
  Arms: bupivacaine

SUMMARY:
To compare the effects of using intrathecal prilocaine combined with fentanyl on duration of motor block versus that of intrathecal bupivacaine combined with fentanyl in elective caesarean section.

DETAILED DESCRIPTION:
The participants in this study will be randomized into two groups based on computer generated numbers using online randomization program (research randomizer). Upon arrival to the operating room, patients will be monitored using electrocardiography, pulse oximetry, and non-invasive blood pressure monitor. The baseline values will be recorded .Heart rate and peripheral oxygen saturation (SpO2) will be monitored continuously; systolic, diastolic, and mean arterial pressure (MAP) will be measured noninvasively at 5 minutes interval during the procedure and during the PACU stay. An 18G-cannulae will be inserted, and pre-medication drugs will be delivered (metoclopramide 10mg). and 4-8 mL/ kg crystalloid infusion will be initiated . Nasal oxygen 3 L / min will be administered during the whole procedure.

* Group P: patients assigned to this group will receive intrathecal 50 mg (2.5 ml) of prilocaine 2% (Takipril, prilocaine hydrochloride 20 mg/mL, hyperbar, Sintetica) + 25 ug fentanyl (0.5 ml).
* Group B: patient assigned to this group will receive intrathecal 10 mg (2 ml) of bupivacaine 5% (sunnypivacaine hyperbaric bupivacaine 20 mg/4ml + 25 ug fentanyl (0.5 ml).

ELIGIBILITY:
Inclusion Criteria:

* Age (18-35)
* ASA II
* Singleton, full term pregnant females.
* Height (1.60-1.90) m.
* BMI > 35 kg m-2
* Scheduled for elective caesarean section under spinal anesthesia.

Exclusion Criteria:

* Patients requiring general anaesthesia
* Known or suspected coagulopathy (international normalised ratio > 1.4), thrombocytopenia (platelet count < 100,000).
* Known peripheral neuropathy, neurological deficits or skeletal deformities.
* Known allergy to prilocaine, bupivacaine , fentanyl.
* Infection at site of injection.
* Patients' refusal to sign informed consent
* Patients with uncontrolled cardiac morbidities (patients with tight valvular lesion, impaired contractility with ejection fraction less than 50%, heart block and arrhythmias), hypertensive disorders of pregnancy, peripartum bleeding.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
time to motor block | time from intrathecal drug injection and time to unassisted ambulation or Bromage's score = 0 (no motor block) (from3 to 5 minutes).

SECONDARY OUTCOMES:
time to sensory block (T4) | time from intrathecal drug injection and complete absence of skin sensation to the pinprick test at T4 (from 1 to 5 minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided